CLINICAL TRIAL: NCT01021371
Title: The GP's Role in Cancer Rehabilitation: a Randomised, Controlled Study.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Vejle Hospital (Other); Vejle Kommune (Unknown)
Responsible Party: Principal Investigator, Stinne Holm Bergholdt, MD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RCT Cancer rehab
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: HRQOL (Health Related Quality Of Life)
Keywords: HRQOL; Rehabilitation; Cancer Patients; General Practice

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient interview and communication to GP from hospital (Experimental): Intervention group: The intervention consists of an extended information routine from hospital to GP based on individual interviews with the patients in the intervention group about their rehabilitation needs and a specific encouragement of the patients' GP to play a proactive role in the patients' rehabilitation course. The individual needs concerning the different types of consequences of the disease and following rehabilitation needs will be brought into focus.
  Interventions: Behavioral: Two step intervention including patient interview followed by an extended information routine to the patients' GP about the patients' rehabilitation needs
- Control group: Usual practice, no intervention (No Intervention)

INTERVENTIONS:
Behavioral: Two step intervention including patient interview followed by an extended information routine to the patients' GP about the patients' rehabilitation needs — The intervention consists of an extended information routine from hospital to GP based on individual interviews with the patients in the intervention group and a specific encouragement of the patients' GP to play a proactive role in the patients' rehabilitation course. The individual needs concerning the different types of consequences of the disease and following rehabilitation needs will be brought into focus. The control group is assigned to usual procedures.
  Arms: Patient interview and communication to GP from hospital

SUMMARY:
The aim of this study is to investigate the impact of a joint effort towards intensifying the collaboration and communication between hospital and general practice.

DETAILED DESCRIPTION:
Background

In recent years an increasing focus has been on the unfulfilled needs of cancer patients for an individual rehabilitation taking into consideration the physical, psychological, social, economic, as well as work-related consequences of the cancer disease. Furthermore, there is a great need for ongoing adjustments of the organisation and procurement of rehabilitation offers and for optimizing the continuity of care, especially regarding transfer between sectors.

Research question

The aim of this study is to investigate whether a joint effort towards intensifying the collaboration and communication between hospital and general practice and encouraging the GP to take an active and prominent part in the rehabilitation process on actual patients has any effect on:

1. Health Related Quality of Life
2. The rehabilitation of cancer patients
3. The experience of continuity of care among cancer patients
4. How the GP act with regard to rehabilitation among cancer patients

Material and methods

The study uses a randomised, controlled design and is carried out as a PhD project. At Vejle Hospital approximately 1000 patients (500 in the intervention group and 500 in the control group) was included at the initiation of treatment. The intervention consists of an extended information routine from hospital to GP based on individual interviews with the patients in the intervention group and a specific encouragement of the patients' GP to play a proactive role in the patients' rehabilitation course. The individual needs concerning the different types of consequences of the disease and following rehabilitation needs will be brought into focus. The data will be obtained from public health registers and questionnaires to patients 6 and 14 months after the time of diagnosis (measuring Health Related Quality of Life, satisfaction with and use of rehabilitation activities, perceived continuity of care and satisfaction with their GP) and to GPs after 12 months (measuring satisfaction with the information from the hospital and activities to meet the patients' rehabilitation needs).

ELIGIBILITY:
Inclusion Criteria:

* All new cancer patients receiving treatment, be it surgery, chemotherapy or radiation, at Vejle Hospital in the period of inclusion.

Exclusion Criteria:

* Patients diagnosed more than 3 months earlier
* Patients younger than 18
* Patients with non-melanoma skin cancer.
* Patients with recurrence of a previous cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | 14 months

SECONDARY OUTCOMES:
How the GP act with regard to rehabilitation among cancer patients | 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Reserch Unit of General Practice, Institute of Public Health, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Bergholdt SH, Hansen DG, Larsen PV, Kragstrup J, Sondergaard J. A randomised controlled trial to improve the role of the general practitioner in cancer rehabilitation: effect on patients' satisfaction with their general practitioners. BMJ Open. 2013 Jul 3;3(7):e002726. doi: 10.1136/bmjopen-2013-002726. Print 2013. PMID 23824312
- [Derived] Bergholdt SH, Larsen PV, Kragstrup J, Sondergaard J, Hansen DG. Enhanced involvement of general practitioners in cancer rehabilitation: a randomised controlled trial. BMJ Open. 2012 Apr 16;2(2):e000764. doi: 10.1136/bmjopen-2011-000764. Print 2012. PMID 22508956